CLINICAL TRIAL: NCT00883519
Title: The Efficacy of Parent Involvement in the Treatment of Adolescent Depression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5758
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Major Depressive Disorder; Dysthymic Disorder; Depressive Disorder NOS; Adjustment Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder; Depression; Adjustment Disorders | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPT-A (Active Comparator)
  Interventions: Behavioral: Interpersonal Psychotherapy for Depressed Adolescents
- IPT-AP (Active Comparator)
  Interventions: Behavioral: Interpersonal Psychotherapy for Depressed Adolescents; Behavioral: Interpersonal Psychotherapy for Depressed Adolescents and Parents

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy for Depressed Adolescents — 12 psychotherapy sessions delivered over 16 weeks
Behavioral: Interpersonal Psychotherapy for Depressed Adolescents and Parents — 12 psychotherapy sessions delivered over 16 weeks
  Arms: IPT-AP

SUMMARY:
The primary aim of this study is to examine whether adolescent depression and the family context in which it develops is best treated using an individual adolescent intervention or an intervention that includes both the adolescent and the parents. This will be accomplished by conducting a randomized controlled pilot study of Interpersonal Psychotherapy for Depressed Adolescents (IPT-A) in comparison to Interpersonal Psychotherapy for Depressed Adolescents and Parents (IPT-AP).

DETAILED DESCRIPTION:
The primary aim of this project is to examine whether adolescent depression and the family context within which it develops is best treated using an individual adolescent intervention or an intervention that includes both the adolescent and the parents. This will be accomplished by conducting a randomized controlled pilot study of Interpersonal Psychotherapy for Depressed Adolescents (IPT-A) in comparison to Interpersonal Psychotherapy for Depressed Adolescents and Parents (IPT-AP). Twenty-two families with adolescents (ages 12-17) who meet criteria for major depressive disorder, dysthymic disorder, depressive disorder NOS, or adjustment disorder with depressed mood and also report elevated levels of parent-adolescent relationship problems will be randomized to receive IPT-A or IPT-AP. Assessments will be administered at screening, baseline, week 4, week 8, week 12, week 16 (post-treatment), and 4 months post-treatment. Outcome measures will include depression symptoms, quality of parent-adolescent relationships, parents' and adolescents' communication skills (assessed through observational coding of a parent-adolescent conflict negotiation task), and adolescents' physiological stress responses to negotiating conflict with a parent (assessed through collection of salivary cortisol). Identifying the best approach to treating both the adolescent's depression and the family environment in which it develops and is maintained would have significant implications for the long-term outcomes of depressed adolescents and their families.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12-17
* English speaking adolescent and parent
* One parent/primary caregiver willing to participate in adolescent's treatment
* Meets diagnostic criteria for Major Depressive Disorder, Dysthymic Disorder, Depressive Disorder NOS, or Adjustment Disorder with Depressed Mood
* BDI-II > 14
* CDRS-R > 36
* CGAS > 65
* CBQ T score >65

Exclusion Criteria:

* Severe episode of Major Depressive Disorder (CDRS-R > 85 and/or PI clinical assessment)
* Current significant risk for suicide (active suicidal ideation with plan; active suicidal ideation without a plan if unable to contract for safety
* Meets diagnostic criteria for substance abuse, schizophrenia, psychosis, bipolar disorder, conduct disorder, or eating disorder
* mental retardation
* medical illness likely to complicate or interfere with treatment
* currently in active treatment for depression
* currently taking medication for a psychiatric diagnosis other than ADHD or not on a stable dose of medication for ADHD (<3 months)
* Parent psychiatrically hospitalized within the past 3 months or parent psychopathology significantly severe to interfere with participation in their adolescent's treatment

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Children's Depression Rating Scale | baseline, week 4, 8, 12, 16, 32

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States